CLINICAL TRIAL: NCT05800262
Title: Dynamic Stability Exercises in Patients With Hypermobile Ehlers-Danlos Syndrome and Hypermobility Spectrum Disorder - a Mixed-methods Feasibility Study
Brief Title: Dynamic Stability Exercises in Patients With Hypermobile Ehlers-Danlos Syndrome and Hypermobility Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Linkoeping University (Other Government); Länssjukhuset i Kalmar län (Other Government); Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Principal Investigator, Helena Romero, Physiotherapist, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1A
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Hypermobility Syndrome; Hypermobile Ehlers-Danlos Syndrome
Keywords: Hypermobility, exercise intervention, feasibility study, EDS
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic stability exercise (Experimental): A dynamic stability exercise program for daily home-exercise was applied during five physiotherapist led sessions distributed over seven weeks.
  Interventions: Behavioral: Dynamic stability exercises

INTERVENTIONS:
Behavioral: Dynamic stability exercises — A dynamic stability exercise program for daily home-exercise was applied during five physiotherapist led sessions distributed over seven weeks.

SUMMARY:
Background:

Symptomatic hypermobility may lead to a number of restrictions in daily life. So far, there is a lack of effective treatments. A whole-body dynamic stability exercise intervention targets to stimulate the dynamic stability and activation of the proprioceptive system and thereby intends to improve patients' health. The aim of the current study was to examine the feasibility, acceptability and impact of a whole-body dynamic stability exercise intervention in patients with hypermobile Ehlers-Danlos syndrome and hypermobility spectrum disorder.

The aim of the current study was to examine the feasibility, acceptability and impact of a dynamic stability exercise intervention in patients with hypermobile Ehlers-Danlos syndrome and hypermobility spectrum disorder.

Methods:

This is a mixed-methods feasibility study. Fifteen patients (14 women and 1 man) with hypermobile Ehlers-Danlos syndrome or hypermobility spectrum disorder and chronic pain were recruited from two pain specialist clinics in the South-East of Sweden. A dynamic stability exercise program for daily home-exercise was applied during five physiotherapist led sessions distributed over seven weeks. Patient reported outcome measures (PROMs) included pain and function, psychological well-being and quality of life. The clinical tests included walking and balance. Through qualitative interviews patients and physiotherapists described their experiences of the assessments and intervention. Assessments were done at baseline, after the intervention, and at the 3-month follow-up.

DETAILED DESCRIPTION:
The specific research questions are:

1. Do retention rates, adherence rates and adverse events allow continuation to a large scale RCT?
2. What are the tendencies of impact of the exercise program on pain, function, psychological well-being and quality of life?
3. Which of the outcome measures used are appropriate and acceptable?
4. What are the patients' and physiotherapists' experiences of the exercise program and protocol.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were adults aged 18 to 67 years old, with generalized hypermobility (castori. A framework), persistent pain (i.e. longer than three months) in at least two of four quadrants of the body and ability to perform the exercises.

Exclusion Criteria:

Exclusion criteria were cancer-related pain, underlying neurological disease, presence of severe psychiatric disorders, known substance abuse, patients in the process of finding optimal medication as well as patients with previous experience of similar exercises.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Identification of suitable measures for a forthcoming RCT | Nine months
  Qualitative and quantitative evaluation through secondaty outcome measures and qualitative interviews with patients and physiotherapists

SECONDARY OUTCOMES:
Pain numeric rating scale | 6 months
  Rating of mean pain last week
Functional Rating Index | 6 months
  Disability regarding daily activities
Multidimensional Fatigue Inventory 20 | 6 months
  Five subscales measuring general fatigue, physical fatigue, reduced motivation, reduced activity and mental fatigue.
  Item 19 was removed according to Hagelin (2009).
Arthritis Self-efficacy scale | 6 months
  Twenty items divided into three sub-scales for self-efficacy for physical function, other symptoms and pain.
Stress and Crisis Inventory-93 | 6 months
  Thirty-five items on physical and psychological symptoms that can be clinical manifestations of stress.
Tampa Scale for Kinesiophobia | 6 months
  Questionnaire measuring kinesiophobia, 17 items.
Orthostatic Hypotension Questionnaire | 6 months
  Assessment of symptoms and daily activity in relation to orthostatic hypotension. 10 items.
European Quality of Life questionnaire (EQ-5D-3L) | 6 months
  Health related quality of life
Berg balance scale | 6 months
  14 tasks common in daily activities testing balance
Bruininks-Oseretsky Test of Motor Proficiency 2 | 6 months
  Nine tasks testing balance
Timed up and go | 6 months
  Mobility, balance, walking ability and fall risk in older adults
2-minute walk test | 6 months
  Walking ability
Wii balance test using a Wii Balance Board | 6 months
  Balance test. Centre of pressure path length, anterio-posterior and medio-lateral sway measured standing on two feet with eyes open and eyes closed, standing on dominant foot and on non-dominant foot with eyes open. Tests performed according to Schmidt (2017), but during 60 seconds instead of 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Romero, Principal Investigator — Smärt- och rehabcentrum, Universitetssjukhuset i Linköping
Locations (2):
- Sweden (2):
  - Samrehab Smärtenheten, the Hospital of Västervik, Västervik, Kalmar County
  - Pain and rehabilitation center, University Hospital of Linkoping., Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Yes
Data is available from the authors on reasonable request.